CLINICAL TRIAL: NCT04053374
Title: Regulation of Lipid Metabolism in Autoimmune Disease: Multiple Sclerosis
Acronym: RELOAD-MS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0057
Record Dates: First submitted 2019-08-05; First posted 2019-08-12 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2019-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample Cerebral Spinal Fluid (CSF) sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- DMD treatment naive CIS or RRMS patients: Newly presenting Clinically Isolated Syndrome (CIS) or Relapsing and Remitting Multiple Sclerosis (RRMS) patients not treated before with Disease Modifying Drugs (DMD) Additional analysis of CSF and CSF cells will be performed in this cohort on a voluntary basis.
  Interventions: Other: Blood sampling
- Secondary Progressive Multiple Sclerosis (SPMS): People with confirmed diagnosis of SPMS
  Interventions: Other: Blood sampling
- Primary Progressive Multiple Sclerosis (PPMS): People with confirmed diagnosis of PPMS
  Interventions: Other: Blood sampling
- DMD-treated with stable disease: People with Multiple Sclerosis (MS) who are treated with DMD who have had stable disease symptoms for at least 3 months
  Interventions: Other: Blood sampling
- Disease controls: People who undergo lumbar puncture due to clinical suspicion of neurological condition, but brain Magnetic Resonance Imaging (MRI) and CSF examination exclude MS diagnosis.
  Interventions: Other: Blood sampling
- Healthy donors: Age, sex and ethnicity matched healthy donors will also be recruited from university and hospital staff and patient friends after informed consent has been obtained. Healthy donors will be asked to provide a blood sample and demographic information but will NOT be asked to provide CSF samples.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling +/- CSF sampling
  Other Names: CSF sampling

SUMMARY:
The aim of this research is to understand how lipids such as cholesterol affect the disease process in people with MS.

DETAILED DESCRIPTION:
In Multiple Sclerosis (MS) immune cells recognise myelin, the coating around nerve fibres, as a foreign molecule and attack it by mistake; at the same time regulatory immune cells (which are normally protective) do not work properly and cannot block the harmful effects of the activated immune cells effectively.

Immune cells work via a complex system of signals that start on the outside layer of the cell (the plasma membrane), these signals are transmitted inside the cell where they trigger immune cell activation. The plasma membrane consists of a fatty layer and changes in the type of fat in the membrane can affect immune cell signalling and immune cell function.

The aims of this project are to:

1. Identify what is different about the types of fat in immune cells from healthy donors and people with MS and identify what triggers the production of these different types of fat.
2. Identify how different types of fat control immune cell function in healthy donors and people with MS
3. Identify possible ways to regulate the type of fat in immune cell membranes to restore normal immune cell function in MS.

Methods: This research study involves collecting participant demographic and clinical information, blood and Cerebral Spinal Fluid (CSF) (optional) from patients with MS. Blood will also be collected from healthy volunteers for comparison. Experiments will be performed on the blood samples and the results correlated with the clinical and disease features of patients.

Outcomes: Many of the molecules involved in the generation of fats are well known and for some of them drugs are already used in humans to treat diseases (for example statins). This could allow the rapid translation of the results from this study to the clinic and have a direct impact for people with MS.

ELIGIBILITY:
Inclusion Criteria:

* 01. Male and female patients of between 18 years and 80 years of age with a diagnosis of MS or CIS.
* Diagnosis confirmed according to the standards at the time when diagnosis was made.
* Patients not receiving biological DMDs within the previous 3 months OR
* Patients treated with DMDs (Interferon beta (Rebif, Betaferon, Avonex, Plegridy), Glatiramer Acetate (Copaxone), Dimethylfumarate (Tecfidera), Fingolimod (Gilenya), Teriflunomide (Aubagio), Natalizumab (Tysabri),) Alemtuzumab (Lemtrada), immunosuppressive drugs (azathioprine, cyclophosphamide etc) who have stable disease in the last 3 months.
* Last course of corticosteroids more than three months ago.
* 02. Having given written informed consent prior to undertaking any study-related procedures.
* 03. Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research.
* 04. Healthy donors ONLY : Male and female donors of between 18 years and 80 years of age in good health and not aware of any diagnosis of an autoimmune condition.

Exclusion Criteria:

* 01. Patients currently taking statins or other lipid lowering therapies.
* 02. Under any administrative or legal supervision.
* 03. Conditions/situations such as:
* Patients with conditions/concomitant diseases making them non evaluable for the primary endpoint
* Impossibility to meet specific protocol requirements (e.g. blood sampling)
* Patient is the Investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Uncooperative or any condition that could make the patient potentially non-compliant to the study procedures
* Pregnant or breast-feeding women, currently or in the last three months prior to inclusion
* Patients who have been vaccinated in the last three months prior to inclusion

Healthy donors ONLY: will be excluded from the study if:

* Donors with a condition likely to influence your blood results such as a current infection or cancer
* Donors who are pregnant or breast-feeding currently or in the last three months
* Donors who have been vaccinated within the last three months
* Donors who cannot provide a blood sample
* Donors who are unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those with and those without MS
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Lipid Phenotyping (1) | 4 hours from point of sample collection
  Blood samples collected from consented participants containing the peripheral blood mononuclear cells (PBMC), serum, Deoxyribonucleic Acid (DNA) and CSF/CSF cells will be appropriately sent to Dr Elizabeth Jury, Centre for Rheumatology Research, University College London (UCL), Rayne Building for lipid phenotyping of PBMC using flow cytometry
Lipid Phenotyping (2) | 4 hours from point of sample collection
  Blood samples collected from consented participants containing the peripheral blood mononuclear cells (PBMC), serum, Deoxyribonucleic Acid (DNA) and CSF/CSF cells will be appropriately sent to Dr Elizabeth Jury, Centre for Rheumatology Research, University College London, Rayne Building for lipid phenotyping of PBMC using measurement of quantitative polymerase chain reaction (qPCR)
Analysis of immune cell function | 4 hours from point of sample collection
  Blood samples collected from consented participants containing the peripheral blood mononuclear cells (PBMC), serum, Deoxyribonucleic Acid (DNA) and CSF/CSF cells will be appropriately sent to Dr Elizabeth Jury, Centre for Rheumatology Research, University College London, Rayne Building for analysis of immune cell function using flow cytometry.
Analysis of cytokine | 4 hours from point of sample collection
  Blood samples collected from consented participants containing the peripheral blood mononuclear cells (PBMC), serum, Deoxyribonucleic Acid (DNA) and CSF/CSF cells will be appropriately sent to Dr Elizabeth Jury, Centre for Rheumatology Research, University College London, Rayne Building for analysis of cytokine using flow cytometry.
Analysis of immune cell function (1) | 4 hours from point of sample collection
  Blood samples collected from consented participants containing the peripheral blood mononuclear cells (PBMC), serum, Deoxyribonucleic Acid (DNA) and CSF/CSF cells will be appropriately sent to Dr Elizabeth Jury, Centre for Rheumatology Research, University College London, Rayne Building for analysis of immune cell function through cell culture.
Analysis of immune cell function (2) | 4 hours from point of sample collection
  Blood samples collected from consented participants containing the peripheral blood mononuclear cells (PBMC), serum, Deoxyribonucleic Acid (DNA) and CSF/CSF cells will be appropriately sent to Dr Elizabeth Jury, Centre for Rheumatology Research, University College London, Rayne Building for analysis of immune cell function through flow cytometry.
Analysis of serum | 4 hours from point of sample collection
  Blood samples collected from consented participants containing serum will be appropriately sent to Dr Elizabeth Jury, Centre for Rheumatology Research, University College London, Rayne Building for measurement of chemokine, lipid expression and expression of other molecules important for immune cell activation.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Farrell, Dr, Principal Investigator — UCL & University College London Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - National Hospital for Neurology and Neurosurgery, London

IPD SHARING:
Plan to Share IPD: Undecided
All participants indicate by written consent if they are willing to allow any of their un-used samples and associated data to be used for future research MS related research.